CLINICAL TRIAL: NCT03067649
Title: Parents' Adherence to Treatment Recommendations: Do It for the Children
Brief Title: Parents' Adherence to Treatment Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12112015113639; U.S. NIH/1RC1MH088329 (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Help-Seeking Behavior
MeSH Terms: conditions — Help-Seeking Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Experimental intervention vs. an information only control
Who Masked: Outcomes Assessor
Masking Description: Evaluators were unaware of condition assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): After the assessment, parents were provided with a 90-minute intervention aimed at increasing the likelihood that the parent would seek treatment for psychiatric problems for themselves.
  Interventions: Behavioral: Motivational Interview
- Information only control (Other): After the assessment, parents were given pamphlet with referral information for psychiatric services.
  Interventions: Behavioral: Information only control

INTERVENTIONS:
Behavioral: Motivational Interview — 90-minute interview to discuss their concerns and possible barriers to seeking treatment for themselves
  Arms: Motivational Interview
Behavioral: Information only control — Participants are provided with a pamphlet containing referral information
  Arms: Information only control

SUMMARY:
The primary purpose of this study was to test whether conducting a brief motivational interview that focused on perceived barriers to treatment seeking would increase the likelihood that a parent with psychiatric problems would seek treatment for themselves.

DETAILED DESCRIPTION:
The primary aim of this study was to test a method for increasing adherence to treatment recommendations for parents of children with emotional/behavior problems. Mental health problems in parents can be a serious risk factor for psychiatric and medical problems in children, yet most parents of children receiving services for mental health or medical problems do not get treatment for their own problems. The specific aim of this study was to increase parents' adherence to recommendations for treatment. Parents were randomly assigned to either the Enhanced Motivational Intervention (EMI) or an information only control group. The EMI involves motivational interviewing comprised of a brief intervention that elicits the parents' "story," provides education about their problem(s), describes the potential link between parents' and children's symptoms, assesses their prior treatment history, expectations, and concerns about treatment, identifies potential barriers to treatment seeking, and determines the next step. Evaluations at baseline and 8-weeks and 4-months post intervention will assess parents' symptoms, functioning, and service utilization. The investigators hypothesized that adherence to treatment recommendations would be significantly greater for parents in the EMI group compared to parents in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of a child who is receiving services for emotional or behavioral problems.
* Must have legal custody of the child

Exclusion Criteria:

* Current psychosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Contact a treatment provider | by the 4-month post intervention evaluation
  Number of participants who contacted a treatment provider

IPD SHARING:
Plan to Share IPD: No
No plan to share the data at this time